











## MEXICAN SOCIAL SECURITY INSTITUTE EDUCATION, RESEARCH AND HEALTH POLICY UNIT HEALTH RESEARCH COORDINATION

HIGH SPECIALTY MEDICAL UNIT (UMAE) "DR. BERNARDO SEPÚLVEDA" CENTRO MÉDICO NACIONAL SIGLO XXI, IMSS, CDMX.

MEDICAL RESEARCH UNIT IN BIOCHEMISTRY.

DEPARTMENT OF NEUROLOGY AND NEUROPHYSIOLOGY.

FAMILY MEDICINE UNITS NUMBER 20, 41 AND 44, IMSS, CDMX. SPECIALTY OF HUMAN ACUPUNCTURE OF THE ENMH OF THE IPN

## Official Title of the study:

"Evaluation of the effect of electroacupuncture on the sensory symptoms of Symmetrical Distal Polyneuropathy of Diabetic origin and its correlation with changes in Nerve Conduction Velocity."

MEXICAN SOCIAL SECURITY INSTITUTE AND EDUCATION, RESEARCH AND HEALTH POLICY UNIT STUDY VERIFICATION ID:

R-2020-785-070.

CONBIOÉTICA-09-CEI-009-20160601.

NCT Number: NOT AVAILABLE.

DOCUMENT OF REAPPROVAL OF THE RESEARCH PROTOCOL.

**DATE:** July 9<sup>th</sup>, 2021.





## Dirección de Prestaciones Médicas

Coordinación de Investigación en Salud División de Desarrollo de la Investigación en Salud Comité de Ética en Investigación



Ciudad de México, a 9 de julio de 2021.

## Dr. José de Jesús Peralta Romero

Investigador Responsable Unidad de Investigación Médica en Bioquímica UMAE, Hospital de Especialidades Centro Médico Nacional Siglo XXI Presente

En relación con el protocolo titulado: "EVALUACIÓN DEL EFECTO DE LA ELECTROACUPUNTURA EN LOS SÍNTOMAS SENSITIVOS DE LA POLINEUROPATÍA DISTAL SIMÉTRICA DE ORIGEN DIABÉTICO Y SU CORRELACIÓN CON CAMBIOS EN LA VELOCIDAD DE CONDUCCIÓN NERVIOSA", con número de registro 2020-785-070, el Comité de Ética en Investigación CONBIOÉTICA-09-CEI-009-20160601 revisó y aprobó la solicitud de reaprobación anual del proyecto por el periodo del 7 de julio de 2021 al 6 de julio de 2022. A su vez, se aprueba el cronograma actualizado.

Sin otro particular, reciba un cordial saludo.

Atentamente

Presidente

Comité de Ética en Investigación

Coordinación de Investigación en Salud

Centro Médico Nacional Siglo XXI